CLINICAL TRIAL: NCT01214434
Title: A Double Blind, Placebo-Controlled, Pilot Study to Estimate the Efficacy and Tolerability of Twice Daily Promiseb Topical Cream in Pediatric Subjects With Cradle Cap (Seborrheic Dermatitis)
Brief Title: Promiseb Topical Cream for Cradle Cap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC0903
Record Dates: First submitted 2010-09-28; First posted 2010-10-05 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Cradle Cap; Infantile Seborrheic Dermatitis
Keywords: Cradle Cap; Infantile seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic; Complement component 5 deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promiseb Topical Cream (Experimental)
  Interventions: Device: Promiseb Topical Cream
- Bland emollient (Sham Comparator)
  Interventions: Other: Bland emollient

INTERVENTIONS:
Device: Promiseb Topical Cream — topical non steroidal cream, twice daily
  Arms: Promiseb Topical Cream
Other: Bland emollient — Eucerin cream twice daily
  Arms: Bland emollient

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Promiseb Topical Cream in cradle cap.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cradle cap
* Must be at least 30 days old
* Must be in good health as determined by investigator
* Naive to prior cradle cap therapy (may have used mineral, olive oils)

Exclusion Criteria:

* Known food, topical product or medicinal allergies.
* Prior use of corticosteroids, antifungals or keratolytics for Cradle Cap
* Weighing less than 7 lbs

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Fraser, PhD, Study Director — Promius Pharma
Locations (4):
- United States (4):
  - Norwich Pediatric Group, Norwich, Connecticut
  - Derm Research, Louisville, Kentucky
  - UMDNJ, Newark, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Bland Emollient: Bland emollient : Eucerin cream twice daily
- Promiseb Topical Cream: Promiseb Topical Cream : topical non steroidal cream, twice daily
Period: Overall Study
Arm/Group | Bland Emollient | Promiseb Topical Cream
Started | 15 | 27
Completed | 11 | 25
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Site error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bland Emollient | Promiseb Topical Cream | Total
Number analyzed (Participants) | 15 | 27 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 27 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.5 (3.5) | 0.8 (1.6) | 1.0 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 6 | 16 | 22
Region of Enrollment [Number; unit: participants]
  United States | 15 | 27 | 42

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Investigator Global Assessment (IGA) Success (IGA of 0 or 1) at End of Treatment (Day 7 or 14).
Description: IGA scored on scale of 0 (clear) to 4 (severe).
Time Frame: end of treatment (Day 7 or 14)
Population: All subjects will data after baseline were included in the analysis. For the Bland emollient group, 2 subjects were excluded from the analysis. For the Promiseb group, 3 subjects were excluded and one of the subjects that did not complete the study was included with Day 7 data carried forward to impute missing Day 14 data.
Measure: Number; unit: percentage of participants
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 13 | 25
percentage of participants | 91.7 | 96
Statistical Analysis 1: Comparison: Bland Emollient vs Promiseb Topical Cream; Test type: Superiority or Other; p > 0.05, Chi-squared

2. Primary Outcome: Number of Participants With Excellent Overall Safety Score at End of Treatment.
Description: The investigator will assess tolerance at Day 7 and Day 14 using an overall safety score of 0 to 3 defined as; Grade 0-No signs of irritation (excellent); Grade 1-Slight signs of irritation which resolved (Good); Grade 2-Clear signs of irritation (Fair); Grade 3-Patient discontinued due to irritation(Poor).
Time Frame: End of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 12 | 25
participants | 12 | 25

3. Secondary Outcome: Precent Reduction From Baseline for Scaling at End of Treatment.
Description: Scaling score on a scale of 0 (none) to 4 (severe).
Time Frame: From Baseline to end of treatment (Day 7 or 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent reduction from baseline
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 12 | 25
percent reduction from baseline | 58 (62) | 90 (22)
Statistical Analysis 1: Comparison: Bland Emollient vs Promiseb Topical Cream; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

4. Secondary Outcome: Percent Reduction From Baseline for Crusting at End of Treatment.
Description: Crusting scored on a scale of 0 (none) to 4 (severe).
Time Frame: From Baseline to end of treatment (Day 7 or 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent reduction from baseline
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 12 | 25
percent reduction from baseline | 85 (22) | 78 (48)
Statistical Analysis 1: Comparison: Bland Emollient vs Promiseb Topical Cream; Test type: Superiority or Other; p = 0.6, t-test, 2 sided

5. Secondary Outcome: Percent Reduction From Baseline for Erythema at End of Treatment.
Description: Erythema scored on scale of 0 (none) to 4 (severe).
Time Frame: From Baseline to end of treatment (Day 7 or 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent reduction from baseline
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 12 | 25
percent reduction from baseline | 74 (43) | 89 (26)
Statistical Analysis 1: Comparison: Bland Emollient vs Promiseb Topical Cream; Test type: Superiority or Other; p = .24, t-test, 2 sided

6. Secondary Outcome: Percent Reduction From Baseline for Oiliness at End of Treatment.
Description: Oiliness scored on a scale of 0 (none) to 4 (severe).
Time Frame: From Baseline to end of treatment (Day 7 or 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent reduction from baseline
Arm/Group | Bland Emollient | Promiseb Topical Cream
Number analyzed (Participants) | 12 | 25
percent reduction from baseline | 88 (23) | 90 (30)
Statistical Analysis 1: Comparison: Bland Emollient vs Promiseb Topical Cream; Test type: Superiority or Other; p = 0.8, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Bland Emollient | Promiseb Topical Cream
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/25
Other Adverse Events (participants affected / at risk) | 1/12 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bland Emollient (N=12) | Promiseb Topical Cream (N=25)
Strep throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects enrolled and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less